CLINICAL TRIAL: NCT00167219
Title: Hematopoietic Cell Transplantation in Children With Juvenile Myelomonocytic Leukemia
Brief Title: Stem Cell Transplant for Juvenile Myelomonocytic Leukemia (JMML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1999LS073; MT1999-20 (Other: Blood and Marrow Transplant Program); 9911M24961 (Other: IRB, University of Minnesota); NCT00262756 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Juvenile Myelomonocytic Leukemia
Keywords: Stem cell transplant; long term survival; retinoic acid
MeSH Terms: conditions — Leukemia, Myelomonocytic, Juvenile | interventions — Stem Cell Transplantation; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intent-to-Treat (Experimental): Patients receiving study regimen.
  Interventions: Biological: Stem Cell Transplant; Drug: Preparative Regimen

INTERVENTIONS:
Biological: Stem Cell Transplant — Transplantation on Day 0.
  Other Names: Bone marrow transplantation
Drug: Preparative Regimen — * Busulfan
  * Cyclophosphamide
  * Mesna
  * Melphalan
  * Anti-thymocyte Globulin (ATG)

SUMMARY:
The investigators hypothesize that long-term disease-free survival (DFS) in patients with JMML can be achieved with a treatment of busulfan (BU), cyclophosphamide (CY) and melphalan (L-PAM) followed by hematopoietic cell transplantation (HCT).

DETAILED DESCRIPTION:
Prior to transplantation, subjects will receive BUSULFAN via the central venous line, six times a day for four days, CYCLOPHOSPHAMIDE via the central venous line once a day for two days, and MELPHALAN via the central venous line for one day. Busulfan, cyclophosphamide, and melphalan are given to destroy the subject's leukemia. As well, these drugs will destroy the subject's own immune system to help ensure the new bone marrow takes and grows after transplantation.

On the day of transplantation, bone marrow or umbilical cord blood from the donor will arrive to the bone marrow transplant unit and be transfused via venous line. These new cells will replace the subject's bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of JMML and fulfill these minimal criteria (International diagnostic criteria for JMML):

  * Leukocytosis (> 13,000) with absolute monocytosis (> 1,000)
  * The presence of immature myeloid cells in the peripheral blood
  * Less than 30% marrow blasts
  * Absence of t(9:22) or BCR-ABL transcript
  * Adequate major organ function including:

    * Cardiac: ejection fraction > 45%
    * Hepatic: no clinical evidence of hepatic failure (e.g. coagulopathy, ascites)
    * Karnofsky performance status > 70% or Lansky score > 50%
    * Creatinine must be < 2 x normal for age
* Written informed consent.

Exclusion Criteria:

* Active uncontrolled infection within one week of HCT.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 1999-11-18 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent-to-Treat: Patients receiving study regimen.
  Stem Cell Transplant: Transplantation on Day 0.
  Preparative Regimen: - Busulfan
  * Cyclophosphamide
  * Mesna
  * Melphalan
  * Anti-thymocyte Globulin (ATG)
Period: Overall Study
Arm/Group | Intent-to-Treat
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Determine Probability of Long-term Disease Free Survival in JMML
Time Frame: at 1 year after transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 15
Percentage of participants | 67 [38 to 85]

2. Secondary Outcome: Combined Incidence of Neutrophil Engraftment, Graft-versus-host Disease (GVHD), Regimen-related Toxicity, and Relapse.
Description: Measured by AGVHD Grades 2 - 4.
Time Frame: at 1 year after transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 15
Percentage of participants | 33 [10 to 57]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intent-to-Treat
All-Cause Mortality (participants affected / at risk) | 4/15
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (N=15)
Aspergillus Fumigatus (Infections and infestations) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hepatomegaly (General disorders) | 2 (5)
Seizure (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (N=15)
Hypertension (Vascular disorders) | 4 (6)
Pericardial Effusion (Cardiac disorders) | 4 (4)
Blood in Stool (Gastrointestinal disorders) | 4 (5)
Blood in Urine (Gastrointestinal disorders) | 1 (1)
Rectal Bleed (Gastrointestinal disorders) | 1 (1)
Bowel Perferation (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Ischemia (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3)
Hickman Line Infection (Infections and infestations) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 4 (5)
Upper respiratory infection (Infections and infestations) | 5 (6)
Lung Infection (Infections and infestations) | 4 (5)
Pneumonia (Reproductive system and breast disorders) | 5 (7)
Dermititis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT00167219/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT00167219/ICF_001.pdf